CLINICAL TRIAL: NCT03750123
Title: Cardiovascular Status of Children 5 Years After Kawasaki Disease
Acronym: CAVASAKI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Principal Investigator, Magdalena Okarska-Napierała, Principal Investigator, Medical University of Warsaw
Other Study IDs: CAVASAKI
Record Dates: First submitted 2018-11-16; First posted 2018-11-21 (Actual); Last update posted 2019-11-25 (Actual); Status verified 2019-11

CONDITIONS: Vasculitis, Systemic; Kawasaki Disease
Keywords: kawasaki; arterial stiffness; PWV; cIMT
MeSH Terms: conditions — Systemic Vasculitis; Mucocutaneous Lymph Node Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples Without DNA — 3 ml of blood will be centrifuged and serum will be stored in separate tubes at - 70°C until analyzed
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Kawasaki Disease (KD): Children 5 years after Kawasaki Disease
- Healthy controls (HC): Age- and sexmatched healthy siblings of children after Kawasaki Disease

SUMMARY:
The aim of present study is to determine cardiovascular status of children who had KD in past and to identify possible biochemical markers of cardiovascular damage in those patients.

In this cross-sectional study children with history of KD will be examined 5 years after receiving intravenous immunoglobulin treatment (IVIG) and compared to healthy controls in terms of: serum levels of endothelial injury markers (circulating endothelial cells, endocan, soluble thrombomodulin, vascular endothelial growth factor (VEGF) and soluble E-selectin), peripheral blood pressure, central blood pressure, arterial stiffness parameters (measured by applanation tonometry), carotid intima media thickness (cIMT), capillaroscopy and echocardiography.

DETAILED DESCRIPTION:
All participants will be examined in Medical University Warsaw Children's Hospital.

Children with history of KD will be recruited from 2 paediatric hospitals in Warsaw and via advertisement by Polish support group for parents of children with KD in social media. Diagnosis of KD will be verified according to current American Heart Association (AHA) guidelines.

All children after KD will be examined 5 years after IVIG treatment exact to 2 months.

CAA presence at the time of KD diagnosis will be determined on the basis of medical records, after specialist consultation, in accordance to AHA definition. Worst-ever echocardiographic picture of coronary arteries will be considered in analysis.

Healthy age- and sex-matched controls (HC) will be recruited from KD patients' siblings.

Informed consent will be obtained from the parents of all patients and all HC.

Assessment of cardiovascular status

All children included in the study will undergo following tests:

1. Laboratory tests

   Blood samples will be drawn after over-night fasting. A) 1.6 ml of blood will be collected in vacutainer tube with ethylenediaminetetraacetic acid (EDTA), B) 4.9 ml of blood will be collected in vacutainer tube with clot-activator, without separation gel (serum tube).

   Routine laboratory techniques will be used to measure lipid profile, glucose and complete blood count. 1 ml of whole blood will be used for circulating endothelial cells (CEC) isolation. CEC will be identiﬁed with CD146-immunomagnetic bead extraction based on an international consensus standardised protocol. 3 ml of blood will be centrifuged at room temperature within 2 h of collection and serum will be stored in separate tubes at -70°C until analyzed. Endothelial injury markers: endocan, soluble thrombomodulin, vascular endothelial growth factor (VEGF) and soluble E-selectin levels will be measured using standardized ELISA assays.
2. Echocardiography

   Echocardiography (ECHO) will be performed with Philips Epiq 7 ultrasound equipment with appropriate transducers by a single specialist supervised by an experienced paediatric echocardiographer. All the standard anatomic and physiological imaging will be done. Multiple imaging planes and transducer positions will be used for optimal visualization of the coronary arteries in all major coronary segments - main stem of left coronary artery, anterior interventricular branch, circumflex branch and right coronary artery will be measured according to AHA guidelines - internal vessel diameter will be assessed from inner edge to inner edge of vessel. The number and location of aneurysms and the presence or absence of intraluminal thrombi and stenotic lesions will be evaluated.

   Another evaluation will include assessment of the left ventricular form and function (ejection fraction measured by Teicholz and Simpson's method, end-systolic and end-diastolic volumes, regional wall motion estimated by M-Mode and speckle tracking modes, evaluation of diastolic function in Tissue Doppler Imaging, both systolic and diastolic function measured as myocardial performance index - i.e. Tei index), aortic root imaging (possible dilatation), valvular function (especially mitral and aortic regurgitation assessed in pulsed and color doppler), presence of pericardial effusion. All of the parameters will be calculated as Z-scores assessed by the health professionals Cardio Z mobile application developed by the experienced Paediatric Cardiology Team at Evelina Children's Hospital in London.
3. Carotid intima media thickness (cIMT)

   cIMT will be evaluated in all subjects by a single experienced specialist using 13-megahertz (MHz) linear transducer, Aloka Prosound Alpha 6, Hitachi Aloka Medical, Mitaka, Japan.

   cIMT will be defined as the mean distance from the leading edge of the lumen-intima interface to the leading edge of the media adventitia interface of the far wall, approximately 1 cm proximal to the carotid bulb. Six determinations of cIMT [mm], three on the left and three on the right side, will be obtained and averaged.
4. Pulse Wave Analysis (PWA) and Pulse Wave Velocity (PWV)

   Arterial pulse waveform and aortal pulse wave velocity will be evaluated by the same investigator using a Sphygmocor device, AtCor Medical Pty Ltd., Sydney, Australia. All pulse wave and velocity measurements will be performed in the sitting position in a quiet, temperature-controlled room (20 ± 5°C) after a 5 min rest.

   Peripheral pressure waveforms will be recorded from the radial artery at the right wrist, using applanation tonometry. After 20 sequential waveforms had been acquired, a validated generalized transfer function will be used to generate the corresponding central aortic pressure waveform.
5. Capillaroscopy

Capillaroscopy will be performed by trained examiner using Dino-Lite Capillaryscope 200 Pro (MEDL4N Pro). The examination will be done in the sitting position, in a temperature-controlled room (20 ± 5°C). The examined finger will be positioned on a base plate and an immersion oil will be applied on the nail fold. Capillary density, morphology and arrangement will be assessed and pictures obtained will be captured and stored through DinoCapture 2.0 software.

All examiners will be unaware of patients' clinical details.

ELIGIBILITY:
Inclusion Criteria:

* history of KD treated with intravenous immunoglobulin (IVIG)

Exclusion Criteria:

* any significant comorbidities,
* body mass index (BMI) value > 1 standard deviation (SD) for age and gender,
* height < 120 cm at the time of cardiovascular assessment.

Ages: 5 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children 5 years after Kawasaki Disease will be recruited from 2 Warsaw hospitals and via advertisment by Polish support group for parents of children with KD in social media
Sampling Method: Non-Probability Sample
Enrollment: 124 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
CEC in children 5 years after KD | 5 years
  comparison of CEC number in KD and HC groups
Arterial stiffness in children 5 years after KD | 5 years
  comparison of pulse wave velocity Z-score in KD and HC groups
Central blood pressure in children 5 years after KD | 5 years
  comparison of central blood pressure values in KD and HC groups

SECONDARY OUTCOMES:
Left ventricle size in children 5 years after KD | 5 years
  comparison of left ventricle mass index in KD and HC groups
Diastolic function of the left ventricle in children 5 years after KD | 5 years
  comparison of E/A ratio in KD and HC groups
cIMT in children 5 years after KD | 5 years
  comparison of cIMT thickness in KD and HC groups
Capillaroscopy in children 5 years after KD | 5 years
  comparison of capillary characteristics (normal / not-normal) in KD and HC groups
Endocan in children 5 years after KD | 5 years
  comparison of endocan serum concentration in KD and HC groups
Thrombomodulin in children 5 years after KD | 5 years
  comparison of thrombomodulin serum concentration in KD and HC groups
VEGF in children 5 years after KD | 5 years
  comparison of VEGF serum concentration in KD and HC groups
Soluble E-selectin in children 5 years after KD | 5 years
  comparison of soluble E-selectin serum concentration in KD and HC groups

CONTACTS AND LOCATIONS:
Overall Officials: Ernest Kuchar, Professor, Study Chair — Medical University of Warsaw
Locations (1):
- Medical University of Warsaw Children's Hospital, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] McCrindle BW, Rowley AH, Newburger JW, Burns JC, Bolger AF, Gewitz M, Baker AL, Jackson MA, Takahashi M, Shah PB, Kobayashi T, Wu MH, Saji TT, Pahl E; American Heart Association Rheumatic Fever, Endocarditis, and Kawasaki Disease Committee of the Council on Cardiovascular Disease in the Young; Council on Cardiovascular and Stroke Nursing; Council on Cardiovascular Surgery and Anesthesia; and Council on Epidemiology and Prevention. Diagnosis, Treatment, and Long-Term Management of Kawasaki Disease: A Scientific Statement for Health Professionals From the American Heart Association. Circulation. 2017 Apr 25;135(17):e927-e999. doi: 10.1161/CIR.0000000000000484. Epub 2017 Mar 29. PMID 28356445
- [Background] Dietz SM, Tacke CE, Hutten BA, Kuijpers TW. Peripheral Endothelial (Dys)Function, Arterial Stiffness and Carotid Intima-Media Thickness in Patients after Kawasaki Disease: A Systematic Review and Meta-Analyses. PLoS One. 2015 Jul 10;10(7):e0130913. doi: 10.1371/journal.pone.0130913. eCollection 2015. PMID 26161871
- [Background] Shah V, Christov G, Mukasa T, Brogan KS, Wade A, Eleftheriou D, Levin M, Tulloh RM, Almeida B, Dillon MJ, Marek J, Klein N, Brogan PA. Cardiovascular status after Kawasaki disease in the UK. Heart. 2015 Oct;101(20):1646-55. doi: 10.1136/heartjnl-2015-307734. Epub 2015 Aug 27. PMID 26316045